CLINICAL TRIAL: NCT03446859
Title: Effect of Transcutaneous Electrical Nerve Stimulation (TENS) on Amelioration of Pain Associated With Primary Dysmenorrhea in Female Undergraduates of a Nigerian University
Brief Title: TENS on Pain Intensity in Primary Dysmenorrhea
Acronym: TENSinPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obafemi Awolowo University (Other)
Responsible Party: Principal Investigator, Adesola Ojo Ojoawo, Dr (Senior Lecturer, Obafemi Awolowo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OJO/2018/001
Record Dates: First submitted 2018-02-19; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Primary Dysmenorrhea
Keywords: Transcutaneous nerve electrical stimulation,; Pain intensity; Primary dysmenorrhea; Female; Undergraduates
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Subjects were randomly allocated to two groups, experimental and control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Experimental): It consists of 25 subjects with primary dysmenorrhea which were put on TENS for 30 minutes, three for 3 days. The subject were placed in supine lying in a comfortable position as possible. The abdomen to the inguinal region were decently exposed and cleaned, after inspection of the area for cuts, skin infections or any abnormalities. A pair of electrodes ( inactive electrodes) will be placed a little below the umbilicus ( Right and Left) and the other pair(active electrode) along the inguinal region at the level of pubic symphysis ( Right and Left) according to (Akinbo et al 2000). A quadripolar method will be used for electrode placement.
  Interventions: Other: TENS
- Control (No Intervention): These are 25 subjects which were not in any intervention. These were subjects that were not placed on TENS and were not used to drug taken for the amelioration of the dysmenorrhea. They were educated on the purpose of research and their inform consent was obtained. Their pain intensity was measured firs, third and 5th days

INTERVENTIONS:
Other: TENS — First, there was explanation of the overall test procedure. The subject was placed in supine lying in a comfortable position.A pair of electrodes (inactive electrodes) was placed a little below the umbilicus (Right and Left) and the other pair (active electrode) along the inguinal region at the level of pubic symphysis (Right and Left) according to (Akinbo et al 2000).
  The TENS equipment was switched on and the intensity was set at a level tolerable by each participant's. The treatment period lasted for 30 minutes for each treatment sessions and the procedure was carried out once a day on the 1st, 3rd and 5th days (Akinbo et.al 2000). Pain intensity was measured pre treatment and post treatment each day of treatment using the visual analogue scale (VAS).
  Other Names: Experimental
  Arms: TENS

SUMMARY:
Dysmenorrhoea is a common problem in women of reproductive age. It is associated with painful uterine contractions and discomfort. The primary aim of the study was to determine the effect of Transcutaneous Electrical Nerve Stimulation (TENS) on pain intensity associated with primary dysmenorrhoea among female undergraduate students of Obafemi Awolowo University.

The study involved 50 females undergraduates of Obafemi Awolowo University with primary dysmenorrhoea lasting for at least 5 days. They were allocated in to two groups equally. One group was treated with TENS and other group served as control. The treatment was for 5 days and Pain intensity was measured before and after the treatment in the two groups. The post treatment pain intensity was then compared.

DETAILED DESCRIPTION:
Subjects

Participants for this study were female undergraduates of OAU presenting with primary dysmenorrhoea.

Sample size determination

Sample size calculation was performed using the following equation: n = (Z2 P (1-P))/(d2), where n = sample size, Z = Z statistic corresponding to a chosen level of confidence, P = expected prevalence, and d = precision. In the calculation; Z will be= 0.9, P= 0.19 and d= 0.05. This calculation will result in a sample size of 50. TENS will be applied for 25 participants and 25 for control.

Sampling technique

A purposive sampling was use to select the Obafemi Awolowo University female students among the undergraduate (participants are volunteers). The consent of the participants were obtained.

Research design It is a true experimental study.

Instrument - Transcutaneous electrical nerve stimulation (MH6000 Combo, MH6100 EMS, MH6200 TENS) manufactured by Medihightec Medical Co., LTD 30175 Hannover, Germany.

* Electrodes (a squared shaped 40 by 40 MM made in the USA).
* Cotton wool
* Methylated Spirit
* Couch
* A Visual Analogue Scale (VAS) (10 Point numerical scale) to rate pain perception of the subjects.

Procedure

Ethical approval was obtained from Health and Ethic Research Committee of Institute of Public Health, Obafemi Awolowo University. Subjects were randomly allocated to two groups. TENS group of 25 and the control of 25. The subjects in the Experimental group was placed in supine lying in a comfortable position as possible. The abdomen to the inguinal region was decently exposed, cleaned using methylated spirit and cotton wool for electrode placement, after inspection of the area for cuts, skin infections or any abnormalities. The absence of such skin conditions as well as intact skin sensation indicates suitability for further procedures. A pair of electrodes ( inactive electrodes) was placed a little below the umbilicus ( Right and Left) and the other pair(active electrode) along the inguinal region at the level of pubic symphysis ( Right and Left) according to. A quadripolar method was used for electrode placement.

Before the commencement of the procedure the subjects was educated about Visual Analogue Scale (VAS).This include how to indicate their pain level. The treatment period lasted for 30 minutes for each treatment sessions and it is once a day for a period of three days that is for the 1st, 3rd and 5th day . The other group did not receive TENS, they served as control. Pain intensity was assessed on the first, 3rd and 5th day from the two groups. Dependent t test was used to compare the mean value of pain intensity within the group on first and 5th day and independent t test was used to compare the mean value of pain intensity on the first day and 5th day between Experimental and control group. Alpha level was set at 0.05

ELIGIBILITY:
Inclusion Criteria:

* Participants with primary dysmenorrhoea, who is single, between the ages of 16 to 30 and have no history of conception, the primary dysmenorrhoea should be at least for five days.

Exclusion Criteria:

* Individuals presenting with pelvic diseases.
* Individuals with cardiac problem.
* Undergraduate with primary dysmenorrhoea but with history of conception.
* Undergraduate with primary dysmenorrhoea currently using analgesia for pain relief.
* Undergraduate with primary dysmenorrhoea not up to five days.

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female undergraduates
Enrollment: 25 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 5 days
  The scale is from 0-5. 0 is no pain 3 is severe pain and 5 is excruciating pain

CONTACTS AND LOCATIONS:
Overall Officials: Adesola O Ojoawo, PhD, Principal Investigator — Obafemi Awolowo University, Ile Ife. Nigeria
Locations (1):
- Obafemi Awolowo University, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Akin M, Price W, Rodriguez G Jr, Erasala G, Hurley G, Smith RP. Continuous, low-level, topical heat wrap therapy as compared to acetaminophen for primary dysmenorrhea. J Reprod Med. 2004 Sep;49(9):739-45. PMID 15493566
- [Result] Adams JM, Taylor AE, Schoenfeld DA, Crowley WF Jr, Hall JE. The midcycle gonadotropin surge in normal women occurs in the face of an unchanging gonadotropin-releasing hormone pulse frequency. J Clin Endocrinol Metab. 1994 Sep;79(3):858-64. doi: 10.1210/jcem.79.3.7521353.